CLINICAL TRIAL: NCT01229592
Title: Clinical Study of Ethanol Lock-therapy in the Prevention of Non-tunnelled, Short Term Central Venous Catheter Associated Infections
Brief Title: Ethanol in the Prevention of Central Venous Catheter Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The non significative reduction of CRBSI adverse events,the need for a high frecuency of catheter manipulations
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC07/90653; 2007-007063-24 (EudraCT Number)
Record Dates: First submitted 2010-10-18; First posted 2010-10-28 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Catheter Related Infection
Keywords: infection; catheter; bacteriaemia; ethanol
MeSH Terms: conditions — Catheter-Related Infections; Infections | interventions — Ethanol; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ethanol (Experimental): Every three day lock using Ethanol in all the lumen of the Catheter
  Interventions: Drug: Ethanol
- Heparine (Active Comparator): Every three day lock using Heparine in all the lumen of the Catheter
  Interventions: Drug: Heparine

INTERVENTIONS:
Drug: Ethanol — Every three day lock using Ethanol(70%)in all the lumen(1ml/per lumen) of the Catheter
  Arms: Ethanol
Drug: Heparine — Every three day lock using Heparin(Fibrilin TM) 3ml in all the lumen of the Catheter
  Arms: Heparine

SUMMARY:
In recent years, several new methods for treatment of catheter-related bloodstream infections (CRBSI) such as antibiotic or antiseptic lock-therapy have been developed with variable success [1-10].

Long-term tunnelled central venous catheters provide a reliable access for administration of chemotherapy, parenteral nutrition or haemodialysis. However, they are not free of complications such as bacteremia. The need to preserve these intra-vascular devices as long as is possible in patients in whom conventional treatment was failed makes emerge antibiotic lock-technique.

Ethanol lock-therapy was demonstrate her utility in this cases. But no study has yet been published using the ethanol lock-therapy as a prophylactic therapy in catheter related infections, neither her application in short-term CVCs.

Objectives: To investigate the value of a ethanol-lock solution in the prophylaxis of non-tunnelled short-term CVC related infections in a heart post-surgical intensive care unit (HPSICU).

Methods: An academic, prospective, randomized and controlled clinical trial is proposed. Patients at HPSICU who have a CVC more than 48 h will be randomized in two arms (ethanol-lock or control group with conventional measurements such as anticoagulants). In the follow-up period, we will register all necessary data to evaluate the end-points of study (CBRSI rate, catheter colonization rate, hospital stay, antimicrobial consume and adverse events due to ethanol).

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* Signed informed consent
* central Venous catheter more than 48 hours placed

Exclusion Criteria:

* pregnancy
* denial Informed consent Form
* ethanol intolerance
* Liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
catheter infectionrelated incidence rates | 2 years
  decrease on catheter infection related incidence rates in comparison to the institution incidence figures

SECONDARY OUTCOMES:
cathether bacteriaemia related rate | 2 years
  versus Institution rate figures
antimicrobial consume | 2 years
  Defined Diary Dosis(DDDs)in both arms

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Microbiología y Enfermedades Infecciosas. Hospital GU Gregorio Marañon, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Perez-Granda MJ, Barrio JM, Munoz P, Hortal J, Rincon C, Rabadan PM, Pernia MS, Bouza E. Ethanol lock therapy (E-Lock) in the prevention of catheter-related bloodstream infections (CR-BSI) after major heart surgery (MHS): a randomized clinical trial. PLoS One. 2014 Mar 27;9(3):e91838. doi: 10.1371/journal.pone.0091838. eCollection 2014. PMID 24675993